CLINICAL TRIAL: NCT01387568
Title: The Effects of Intravenous Lidocaine Infusion During and After Major Abdominal Pediatric Surgery. A Randomized Double-blinded Study
Brief Title: Lidocaine Infusion for Major Abdominal Pediatric Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Associate Professor of Anesthesiology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MUH-AD-1-2011
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Elective Major Abdominal Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group L (Active Comparator): Lidocaine group
  Interventions: Drug: Lidocaine Infusion
- group P (Placebo Comparator): Placebo group
  Interventions: Drug: saline Infusion

INTERVENTIONS:
Drug: Lidocaine Infusion — children in group L received i.v. lidocaine 1.5 mg/kg followed by infusion at 1.5 mg. kg-1.h-1. and were continued up to 6 hours postoperatively
  Arms: group L
Drug: saline Infusion — children in group P received i.v. saline 0.9% 1 ml/kg followed by infusion at 0.1 ml. kg-1.h-1,and were continued up to 6 hours postoperatively
  Arms: group P

SUMMARY:
In this study, the investigators hypothesized that perioperative i.v. infusion of lidocaine in major abdominal pediatric surgery, may have a beneficial effect on hemodynamic and hormonal responses. Also, it could decrease the hospital stay, opioid requirement and hasten return of bowel function.

DETAILED DESCRIPTION:
The inflammatory response after major abdominal surgery is of great importance for patients, physicians and perioperative medicine1. Perioperative excessive stimulation of the inflammatory and hemostatic systems may result in development of postoperative ileus, ischemia-reperfusion syndromes, hypercoagulation syndromes (e.g. deep venous thrombosis) and pain excessive inflammatory response such as impaired gastrointestinal motility, so modulation of inflammatory responses may decrease severity of such complications 2,3.

Intravenous lidocaine, a local anesthetic, has been shown to improve postoperative analgesia, reduce postoperative opioid requirements, accelerate postoperative recovery of bowel function, attenuate postoperative fatigue, reduced the duration of hospitalization, and facilitate acute rehabilitation in patients undergoing laparoscopic abdominal surgery 4. Administration of local anesthetics to epidural space has analgesic effect, blunt stress response; provide rapid mobilization, early extubation with rapid recovery of bowel function 5. However, insertion of an epidural catheter carries risks especially in pediatric populations. So, systemic lidocaine may become another strategy for improving perioperative outcome which is safe and effective2.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric
* Abdominal surgery
* ASA class I and II

Exclusion Criteria:

* history of hepatic diseases
* history of cardiac diseases
* history of renal diseases
* allergy to local anesthetics
* epilepsy

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure | for 2hrs after infusion

SECONDARY OUTCOMES:
Plasma Cortisol | for 24 hrs after infusion
Serum lidocaine | 6 hrs after infusion
  The TDx/ TDx FLx (Abbot Diagnostic, USA) lidocaine assay was used for quantitative measurement of serum lidocaine
Heart rate (HR) | for 6 hrs after infusion
Pain scales | 24 hrs postoperative
  In the postanaesthetic care unit (PACU), children were assessed for pain every 10 min by the trained nurse blinded to group assignment, using 1 of 2 pain scales according to child comprehension: a 0- to 10-point visual analog scale (VAS), or FLACC Scale (Face, Legs,Activity, Cry, Consolability). FLACC is an observer assessment based 5 items and each item is graded from 0 to 2

CONTACTS AND LOCATIONS:
Overall Officials: Alaa El Deep, MD, Principal Investigator — alaaeldeep9@hotmail.com
Locations (1):
- Anesthesia Dept, Mansoura University, Al Mansurah, DK, Egypt